CLINICAL TRIAL: NCT00271986
Title: Intraperitoneal Microdialysis Monitoring of Patients During the Early Postoperative Period After LAR With Reference to Early Diagnosis of Anastomotic Leakage
Brief Title: Peritoneal Microdialysis in Patients Undergoing Low Anterior Resection (LAR) for Recto-sigmoid Cancer
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Niels Qvist, professor, Niels Qvist, Professor, Surgical Department A, Odense Universityt Hospital
Other Study IDs: VF20050008
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2008-05

CONDITIONS: Cancer of Rectum
Keywords: Peritoneal microdialysis; Low anterior resection; Recto-sigmoid cancer; Anastomotic leakage
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Anastomotic leakage is a serious complication after LAR with high morbidity and mortality rates. Early diagnosis and treatment is mandatory. The primary aim of the present study is to investigate the clinical use of peritoneal microdialysis and whether is able to detect anastomotic leakage prior to clinical symptoms develops.

DETAILED DESCRIPTION:
Patients undergoing LAR for recto-sigmoid cancer is subjected to peritoneal microdialyses during the postoperative period until discharge. Subcutaneous microdialysis serve as control. Samples are collected every 4-hour. Samples will be analyzed continuously but the results will not be included in the clinical evaluation of the patient.

Patients undergoing abdomino-perineal rectal resection will serve as a control group.

A total of 50 patients will be included in this pilot study. The results of the peritoneal microdialyses will be compared with the clinical course in each patient. The results form the uncomplicated courses will be used to define the normal variations in peritoneal microdialysis. This will be compared to results from patients with various complications.

The study is approved by the local scientific ethical committee No. ------

ELIGIBILITY:
Inclusion Criteria:

* Histological verified cancer
* The cancer must be located in rectum or the sigmoid colon
* Diverting stoma is allowed
* Perioperative radio-chemotherapy is allowed

Exclusion Criteria:

* Disseminated cancer
* ASA-group 4 ore higher

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing Loa Anterior Resection (LAR) or rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
anastomotic leakage | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Niels Qvist, Professor, Study Chair — Odense University Hospital
Locations (1):
- Deparment A, Odense, Denmark